CLINICAL TRIAL: NCT00747188
Title: The Impact of Problem-Based Learning (PBL) and Lecturing on the Behavior and Attitudes of Iranian Nursing Students: a Randomised Controlled Trial (RCT)
Brief Title: The Impact of Problem-Based Learning (PBL) and Lecturing
Acronym: PBL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tasmania (Other)
Responsible Party: Dr Heydarnejad, Assistant Professor
Purpose: Health Services Research
Other Study IDs: SAEED1
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Last update posted 2008-09-04 (Estimated); Status verified 2008-09

CONDITIONS: Learning
Keywords: Problem-based learning (PBL); lecture; nursing; education; none of students had any prior exposure to PBL

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Experimental)
  Interventions: Behavioral: PBL
- A, 2, III (No Intervention)

INTERVENTIONS:
Behavioral: PBL
  Arms: 2

SUMMARY:
The present study aimed to compare the effect of education through problem-based learning (PBL) or lectures on behavior, attitude and learning of nursing students.

DETAILED DESCRIPTION:
A total of 40 second-year nursing students participated: 20 students in the PBL group and 20 students in the traditional lecture (control) group. The students underwent a one-semester course using the two methods of education

ELIGIBILITY:
Inclusion Criteria:

* Students must not have been exposed to PBL

Exclusion Criteria:

* Biased and specific students

Ages: 19 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2006-02; Primary Completion 2007-07 (Actual); Study Completion 2008-01 (Actual)

REFERENCES:
- [Derived] Dehkordi AH, Heydarnejad MS. The impact of problem-based learning and lecturing on the behavior and attitudes of Iranian nursing students. A randomised controlled trial. Dan Med Bull. 2008 Nov;55(4):224-6. PMID 19232163